CLINICAL TRIAL: NCT02034383
Title: Macronutrient Absorption From Almonds: The Effect of Processing on the Measured Energy Value of Almonds in the Human Diet
Brief Title: The Effect of Processing on the Measured Energy Value of Almonds in the Human Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Baer (U.S. Federal Agency)
Collaborators: Almond Board of California (Other)
Responsible Party: Sponsor-Investigator, David Baer, Research Physiologist, USDA Beltsville Human Nutrition Research Center
Organization: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: HS45
Record Dates: First submitted 2014-01-09; First posted 2014-01-13 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Healthy; Focus: Effect of Processing on Energy Value of Almonds

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Control (Experimental): Diet will consist of a controlled diet without almonds for 3 weeks.
  Interventions: Other: Control
- Whole Almonds (Experimental): Diet will consist of a controlled diet with whole almonds for 3 weeks.
  Interventions: Other: Whole Almonds
- Roasted Whole Almonds (Experimental): Diet will consist of a controlled diet with roasted whole almonds for 3 weeks.
  Interventions: Other: Roasted Whole Almonds
- Diced Almonds (Experimental): Diet will consist of a controlled diet with diced almonds for 3 weeks.
  Interventions: Other: Diced Almonds
- Almond Butter (Experimental): Diet will consist of a controlled diet with almond butter for 3 weeks.
  Interventions: Other: Almond Butter

INTERVENTIONS:
Other: Control — Controlled diet for 3 weeks with 0 servings/day of almonds.
  Arms: Control
Other: Whole Almonds — Controlled diet for 3 weeks with 1.5 servings/day of whole, natural almonds.
  Arms: Whole Almonds
Other: Roasted Whole Almonds — Controlled diet for 3 weeks with 1.5 servings/day of roasted whole almonds.
  Arms: Roasted Whole Almonds
Other: Diced Almonds — Controlled diet for 3 weeks with 1.5 servings/day of diced almonds.
  Arms: Diced Almonds
Other: Almond Butter — Controlled diet for 3 weeks with 1.5 servings/day of almond butter.
  Arms: Almond Butter

SUMMARY:
The objective of this study is to measure the effect of processing (roasting, slicing, or grinding) on the energy value of almonds in the human diet and study molecular mechanisms that may help explain the beneficial health effects of almonds.

DETAILED DESCRIPTION:
The metabolizable energy values, or Atwater general factors, for protein, fat, and carbohydrate are commonly used to calculate the metabolizable energy of a diet. Atwater factors are based on average values of mixed diets and are not exact; thus, using these values could introduce an error in the calculated metabolizable energy of a particular food due to differences in chemical structure and availability. Studies have demonstrated that Atwater general factors overestimate the energy derived from protein and fat, as well as the measured metabolizable energy of mixed diets, particularly those that are high in dietary fiber. Studies are lacking, however, that examine how different processing methods affect the metabolizable energy of a food due to differences in chemical structure and availability.

ELIGIBILITY:
Inclusion Criteria:

* Age 25 to 75 years at beginning of study
* BMI between 20 and 38 kg/m2
* Fasting glucose < 126 mg/dl
* Blood pressure < 160/100 (controlled with certain medications)
* Fasting total blood cholesterol < 280 mg/dl
* Fasting triglycerides < 300 mg/dl

Exclusion Criteria:

* Presence of kidney disease, liver disease, gout, hyperthyroidism, untreated or unstable hypothyroidism, certain cancers, gastrointestinal disease, pancreatic disease, other metabolic diseases, or malabsorption syndromes
* Women who have given birth during the previous 12 months
* Pregnant women or women who plan to become pregnant or become pregnant during the study
* Lactating women
* Type 2 diabetes requiring the use of oral antidiabetic agents or insulin
* History of bariatric or certain other surgeries related to weight control
* Smokers or other tobacco users (during 6 months prior to the start of the study)
* History of eating disorders or other dietary patterns which are not consistent with the dietary intervention (e.g., vegetarians, very low fat diets, high protein diets)
* Volunteers who have lost 10% of body weight within the last 12 months
* Known (self-reported) allergy or adverse reaction to almonds or other nuts
* Unable or unwilling to give informed consent or communicate with study staff
* Self-report of alcohol or substance abuse within the past 12 months and/or current acute treatment or rehabilitation program for these problems (long-term participation in Alcoholics Anonymous is not an exclusion)
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Metabolizable Energy | End of each 3-week diet period
  The metabolizable energy value of almonds and almond butter will be calculated based on the chemical composition and energy content of the consumed diet and excreta.

SECONDARY OUTCOMES:
Digestibility | End of each 3-week diet period
  Fat, protein, and fiber digestibility will be calculated and the effect of almond on nutrient digestibility will be assessed.
Almond nutrient metabolism | End of each 3-week diet period
  Blood and urine will be analyzed for appearance of almond nutrients and their metabolites.
Biomarkers of cardiovascular disease | End of each 3-week diet period
  Blood will be analyzed for biomarkers of risk for cardiovascular disease and cancer such as oxidative stress and inflammatory markers.

CONTACTS AND LOCATIONS:
Overall Officials: David J. Baer, Ph.D., Principal Investigator — USDA Beltsville Human Nutrition Research Center
Locations (1):
- USDA Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States

REFERENCES:
- [Background] Novotny JA, Gebauer SK, Baer DJ. Discrepancy between the Atwater factor predicted and empirically measured energy values of almonds in human diets. Am J Clin Nutr. 2012 Aug;96(2):296-301. doi: 10.3945/ajcn.112.035782. Epub 2012 Jul 3. PMID 22760558